CLINICAL TRIAL: NCT05776589
Title: The Effect of Pressure Controlled Volume Guaranteed Ventilation and Volume Controlled Ventilation on Hemodynamics and Lung Dynamics in Prone Position Patients in Thoracolomber Vertebra Surgery
Brief Title: The Effect of Intraoperative Ventilation Mode on Hemodynamics and Lung Dynamics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Arslan Yurtlu, Associate Professor, Izmir Ataturk Training and Research Hospital
Other Study IDs: Izmir ATRH
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation
Keywords: lung dynamics under general anesthesia; prone position; pressure controlled mode; volume controlled mode; vertabral surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group PCV-VG: In this group, pressure-controlled volume guaranteed ventilation (PCV- VG) was applied in patients undergoing vertebral surgery in the prone position.
  Interventions: Device: The mechanical ventilation mode
- Group VCV: In this group, volume-controlled ventilation (VCV) was applied in patients undergoing vertebral surgery in the prone position.
  Interventions: Device: The mechanical ventilation mode

INTERVENTIONS:
Device: The mechanical ventilation mode — Changing the mechanical ventilation mode

SUMMARY:
In this study, it was aimed to compare the effects of pressure-controlled volume-guaranteed ventilation (PCV-VG) and volume-controlled ventilation (VCV) on lung dynamics and hemodynamics in patients undergoing vertebral surgery in the prone position.

DETAILED DESCRIPTION:
The VCV (volume controlled ventilation) mode is the mode commonly used in general anesthesia practice. In VCV mode, the parameters under control are tidal volume and respiratory rate. In VCV mode, airway pressure changes depending on resistance and compliance. There is a risk of increased airway pressures in this mode.

In PCV-VG (pressure controlled volume guaranteed ventilation) mode, the parameters under control are the peak airway inspiratory pressure and the I/E ratio. It has been shown that peak airway pressures decrease and partial oxygen pressure increase due to decreased inspiratory flow in this ventilation mode.

Both ventilation modes are frequently used in patients undergoing general anesthesia.

In this study, it was aimed to compare the effects of pressure-controlled volume-guaranteed ventilation (PCV-VG) and volume-controlled ventilation (VCV) on lung dynamics (pulmonary peak-plateau pressure, compliance, driving pressure, SpO2 and end-tidal carbon dioxide) and hemodynamics (mean arterial pressure and heart rate) in patients undergoing vertebral surgery in the prone position.

In the study, patients will be randomized and divided into 2 groups after obtaining informed consent forms. If a mode change is required during the surgery, that patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo thoracolumbar vertebral surgery in the prone position
* Patients older than 18 years
* Patients younger than 70 years of age
* ASA 1-2 patients

Exclusion Criteria:

* Patients with a BMI >30 kg/m2
* Patients with a history of chronic pulmonary disease
* Patients with a history of previous thoracic surgery
* Patients with ASA >3
* Patients who will undergo emergency surgery
* Pregnant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vertebral surgery in the prone position.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effects of pressure controlled volume guaranteed ventilation and volume controlled ventilation on lung compliance | 3 months
  Comparison of the effects of pressure controlled volume guaranteed ventilation (PCV-VG) and volume controlled ventilation (VCV) on lung compliance (ml/cmH20) in patients undergoing vertebral surgery in a prone position

SECONDARY OUTCOMES:
Comparison of the effects of pressure controlled volume guaranteed ventilation and volume controlled ventilation on heart rate | 3 months
  Comparison of the effects of pressure controlled volume guaranteed ventilation (PCV-VG) and volume controlled ventilation (VCV) on heart beats per minute (bpm) in patients undergoing vertebral surgery in a prone position
Comparison of the effects of pressure-controlled volume guaranteed ventilation and volume-controlled ventilation on mean arterial pressure | 3 months
  Comparison of the effects of pressure controlled volume guaranteed ventilation (PCV-VG) and volume controlled ventilation (VCV) on mean arterial pressure (mmHg) in patients undergoing vertebral surgery in a prone position

CONTACTS AND LOCATIONS:
Overall Officials: Derya A Yurtlu, M.D., Principal Investigator — Izmir Atatürk Training and Reseach Hospital
Locations (1):
- KCU Izmir Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No